CLINICAL TRIAL: NCT00703066
Title: A Phase I, Randomized, Controlled, Double-Blind, Single Centre Trial to Evaluate the Safety and Immunogenicity of 30 and 100 µg of GMZ2 in Gabonese Children Aged 1-5 Years
Brief Title: Safety and Immunogenicity of 30 and 100 µg of GMZ2 in Gabonese Children Aged 1-5 Years
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: African Malaria Network Trust (Network)
Responsible Party: Roma Chilengi, African Malaria Network Trust
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GMZ2_3_08
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: Malaria
Keywords: Malaria; Vaccine; GMZ2; Safety; African; immunogenicity
MeSH Terms: conditions — Malaria | interventions — Rabies Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): three doses of 30µg GMZ2,
  Interventions: Biological: GMZ 2 vaccine (GLURP + MSP 3)
- 2 (Experimental): 3 doses of 100 µg of GMZ2
  Interventions: Biological: GMZ 2 vaccine (GLURP + MSP 3)
- 3 (Active Comparator): Rabies vaccine
  Interventions: Biological: Rabies vaccine

INTERVENTIONS:
Biological: GMZ 2 vaccine (GLURP + MSP 3) — three doses of 30µg of GMZ 2 vaccine,
  Arms: 1
Biological: GMZ 2 vaccine (GLURP + MSP 3) — 100 µg of GMZ 2 vaccine
  Arms: 2
Biological: Rabies vaccine — 3 doses of Rabies vaccine
  Arms: 3

SUMMARY:
The study aims to show that the candidate malaria vaccine GMZ2 is as safe as the already publicly used vaccine against rabies. 30 Gabonese children aged 1-5 years will be enrolled and randomly allocated to receive either malaria vaccine or rabies vaccine without the investigator or the participants knowing what they received. They will receive 3 doses each at one month intervals, and will be followed up for one year to evaluate safety parameters. 30 and 100µg doses for the candidate malaria vaccine GMZ 2 will be evaluated for safety.

This is the second time that candidate malaria vaccine GMZ 2 is being tested in Africa, the first time being in Gabonese adults where the product was found to be safe.

DETAILED DESCRIPTION:
Background. GMZ2 is a recombinant hybrid of the Glutamate Rich Protein (GLURP) and the Merozoite Surface Protein 3 (MSP 3).This product has been developed at State Serum Institute/EMVI in Denmark and Batch released by Henogen of Belgium. The phase Ia trial in malaria naive volunteers was done in Germany, at Tuebingen University. This phase Ia trial established safety of the vaccine and also assisted in selecting the best dosage (10, 30 or 100 µg). The dosage with the best safety and immunogenicity profile will be tested for the phase Ib trials in Gabon, including this phase Ib trial in children.

Objectives:

Primary objective:

To evaluate the safety and reactogenicity of three doses of 30 and 100µg GMZ2, adsorbed on aluminium hydroxide, in comparison with three doses of the control vaccine (rabies), in healthy Gabonese children aged 1-5 years.

Secondary objectives:

To assess the humoral immune response to the vaccine antigens GMZ2, GLURP and MSP3 by measuring the total IgG concentration and IgG isotypes against GMZ2 by ELISA.

To assess B-cell memory by memory B-cell ELISPOT.

Exploratory Objectives:

To assess the functionality of the immune response by measuring the Growth Inhibition of P. falciparum in the presence or absence of Monocytes, and by measuring the recognition of native antigen of P. falciparum by IFA.

Study Design:

Phase Ib double-blind, randomised, and controlled trial with three groups at one study site; rabies vaccine,30µg and 100 µg GMZ 2 vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Children age 1-5 years inclusive at the time of screening;
* Residing in Lambaréné for the duration of the study;
* Written informed consent obtained before screening and study start, respectively;
* Available to participate in follow-up for the duration of study (13 months);
* General good health based on history and clinical examination.

Exclusion Criteria:

* Previous vaccination with any other malaria candidate vaccine.
* Concomitant vaccination with a investigational vaccine or a rabies vaccine;
* Use of a investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first study vaccination, or planned use up to 30 days after the third vaccination;
* Chronic administration (defined as more than 14 days) of immuno-suppressants or other immune-modifying drugs within six months prior to the first vaccination. This includes any dose level of oral steroids or inhaled steroids, but not topical steroids;
* Confirmed or suspected immunosuppressive or immuno-deficient condition, including human immunodeficiency virus (HIV) infection;
* Confirmed or suspected autoimmune disease;
* History of allergic reactions or anaphylaxis to immunizations or to any of the vaccine components, or of serious allergic reactions to any substance, requiring hospitalization or emergent medical care;
* History of splenectomy;
* Laboratory evidence of liver disease (Alanine aminotransferase [ALT] greater than 1.25 times the upper limit of normal (<45 U/L) of the testing laboratory);
* Laboratory evidence of renal disease (serum creatinine greater than the upper limit of normal of the testing laboratory, or more than trace protein or blood on urine dipstick testing);
* Laboratory evidence of haematological disease (absolute leukocyte count 3.5-11/µL, absolute lymphocyte count 560-5280/µL, platelet count 120,000-400,000/µL, or haemoglobin 10.0-16.5g/dL);
* Administration of immunoglobulins and/or any blood products within the three months preceding the first study vaccination or planned administration during the study period;
* Simultaneous participation in any other interventional clinical trial;
* Acute or chronic pulmonary, cardiovascular, hepatic, renal or neurological condition, malnutrition, or any other clinical findings that in the opinion of the clinical investigator, may increase the risk of participating in the study;
* Other condition that in the opinion of the clinical investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-07 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Immediate reactogenicity. | within 30 minutes after each injection
Local and systemic reactogenicity | 14 days following each immunization
unsolicited Adverse events | up to 1 month after the 3rd vaccination
Occurrence of serious adverse events | 1 year
Biological safety | 1 year

SECONDARY OUTCOMES:
Humoral immune response to GLURP and MSP 3 | 1 year
Cellular immune response | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kremsner, MD, PhD, Study Director — Medical research Unit, Albert Schweitzer Hospital
Locations (1):
- Medical Research Unit, Albert Schweitzer Hospital, Lambaréné, Gabon

REFERENCES:
- [Derived] Belard S, Issifou S, Hounkpatin AB, Schaumburg F, Ngoa UA, Esen M, Fendel R, de Salazar PM, Murbeth RE, Milligan P, Imbault N, Imoukhuede EB, Theisen M, Jepsen S, Noor RA, Okech B, Kremsner PG, Mordmuller B. A randomized controlled phase Ib trial of the malaria vaccine candidate GMZ2 in African children. PLoS One. 2011;6(7):e22525. doi: 10.1371/journal.pone.0022525. Epub 2011 Jul 28. PMID 21829466